CLINICAL TRIAL: NCT06917885
Title: Phase Ib Open-label Study of Adjuvant CUE-102, a WT-1-pHLA-IL2-Fc Fusion Protein in Glioblastoma (GBM) Patients at First Recurrence
Brief Title: CUE-102 in Recurrent Glioblastoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: David Reardon, MD (Other)
Collaborators: Cue Biopharma (Industry)
Responsible Party: Sponsor-Investigator, David Reardon, MD, Sponsor-Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-023
Record Dates: First submitted 2025-04-07; First posted 2025-04-09 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Glioblastoma; Glioblastoma; Glioma, Malignant
Keywords: Glioblastoma; Recurrent Glioblastoma; Glioma, Malignant
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CUE-102 (Experimental): The first 12 participants will be enrolled using a standard 3 + 3 design in a safety lead-in to determine the maximum tolerated dose (MTD) of CUE-102 per protocol. Once the MTD has been determined, up to 6 additional participants will be enrolled in a dose expansion cohort. Participants will complete:
  * Baseline visit
  * Imaging every 9 weeks starting at Cycle 3
  * Cycle 1 through End of Treatment (up to 1 year in total, approximately 17 cycles)
    --Day 1 of 21 day cycle: Predetermined dose of CUE-102 1x daily.
  * End of Treatment visit with imaging
  * Long-Term Follow Up: every 3-4 months
  Interventions: Biological: CUE-102

INTERVENTIONS:
Biological: CUE-102 — A WT-1-pHLA-IL2-Fc fusion protein, single-use vial, via intravenous (into the vein) infusion per protocol.

SUMMARY:
The goal of this study is to evaluate the safety of the experimental drug, CUE-102, and establish the recommended dose of CUE-102 for participants with Recurrent Glioblastoma (GBM).

The name of the study drug involved in this study is:

-CUE-102 (a type of fusion protein)

DETAILED DESCRIPTION:
This is a single center, open-label, Phase Ib trial evaluating the safety and tolerability of CUE-102 monotherapy in adult participants with Glioblastoma (GBM) at first recurrence. CUE-102 is designed to target tumor cells by activating T cells, potentially improving clinical outcomes in recurrent GBM.

The U.S. Food and Drug Administration (FDA) has not approved CUE-102 as a treatment for Recurrent Glioblastoma.

The research study procedures include screening for eligibility, in-clinic visits, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, blood and urine tests, and electrocardiograms (ECG).

It is expected that about 18 people will take part in this research study.

Cue Biopharma, Inc. is supporting this research study by providing the study drug, CUE-102.

ELIGIBILITY:
Inclusion Criteria:

* Have HLA-A*0201 genotype as determined by genomic testing performed locally;
* Have histologically confirmed World Health Organization (WHO) Grade 4 glioblastoma, other WHO grade 4 malignant glioma or molecular GBM (based on the 2021 WHO Classification) at first recurrence. Patients with gliosarcoma are NOT eligible;
* Be willing and able to provide written informed consent/assent for the trial;
* Be ≥ 18 years of age on day of signing informed consent;
* Have a Karnofsky performance status (KPS) ≥ 70 (Appendix A);
* Participants must be at least 4 weeks from start of last chemotherapy cycle (at least 6 weeks for nitrosoureas and at least 1 week for metronomic dosing) and at least 4 weeks or 5 half-lives (whichever is shorter) for any prior investigational agent. There is no minimal time from cessation of Optune TTF nor for prior cancer vaccine therapy.
* MRI within 14 days prior to registration. MRIs should include vascular imaging when possible. Corticosteroid dose must be stable or decreasing for at least 5 days prior to the scan. If steroids are added or the steroid dose is increased between the date of the screening MRI scan and the start of treatment, a new baseline MRI or CT is required;
* Patients must have fully completed initial radiation therapy with or without daily temozolomide including 60 Gy in 30 fractions, 59.4 Gy in 1.8 Gy per fraction or equivalent;
* At least 12 weeks from completion of radiotherapy +/- temozolomide. Patients < 12 weeks from the completion of radiation therapy may be eligible if they have either of the following: 1) histopathologic confirmation of recurrent tumor; or 2) new contrast enhancing disease outside the primary radiation field. Participants who have received investigational therapies as a component of treatment for newly diagnosed GBM as long as remaining eligibility criteria are satisfied;
* Participants must have recovered to grade 0 or 1 or pre-treatment baseline from clinically significant toxic effects of prior therapy (exceptions include alopecia, laboratory values listed per inclusion criteria, and lymphopenia, which is common after therapy with temozolomide);
* Participants must meet the following organ and marrow function as defined below, all screening labs should be performed within 14 days of registration:

  * Absolute neutrophil count (ANC) ≥1,500 /mcL
  * Platelets ≥100,000 / mcL
  * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L (Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks)
  * Serum creatinine ≤ 1.5 X institutional ULN OR
  * Measured or calculated creatinine clearance (CrCl) ≥45 mL/min for participant with creatinine levels > 1.5 X institutional ULN (CrCl should be calculated per institutional standard, GFR can also be used in place of creatinine or CrCl)
  * Serum total bilirubin ≤ 1.5 X institutional ULN OR
  * Direct bilirubin ≤ institutional ULN for participants with total bilirubin levels > 1.5 X institutional ULN
  * AST (SGOT) and ALT (SGPT) ≤ 3.0 X institutional ULN OR ≤ 5 X institutional ULN for participants with Gilberts syndrome
  * International Normalized Ratio (INR) OR Prothrombin Time (PT) and Activated Partial Thromboplastin Time (aPTT) ≤1.5 X institutional ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
  * Resting baseline oxygen saturation by pulse oximetry ≥92% at rest
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must have a negative urine or serum pregnancy within 72 hours prior to enrollment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required;

  --Women in the following categories are not considered WOCBP:
  * Premenarchal
  * Premenopausal female with 1 of the following:

    * Documented hysterectomy
    * Documented bilateral salpingectomy
    * Documented bilateral oophorectomy
    * Note: Documentation can come from the site personnel's review of the participant's medical records, medical examination, or medical history interview.
  * Postmenopausal female

    * A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.

      -----A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy (HRT). However, in the absence of 12 months of amenorrhea, confirmation with two FSH measurements in the postmenopausal range is required.
    * Females on HRT and whose menopausal status is in doubt will be required to use one of the non-hormonal highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before study enrollment.
* Women of child-bearing potential (WOCBP; see definition above), must agree to use a highly effective method of contraception consistently and correctly as described below during study treatment and for 120 days after study treatment discontinuation or the initiation of other cancer therapy (whichever is shorter);

  * Highly Effective Contraceptive Methods That Are User Dependent a (Failure rate of < 1% per year when used consistently and correctly.)
  * Combined (estrogen- and progestogen- containing) hormonal contraception

    * i. Oral
    * ii. Intravaginal
    * iii. Transdermal
    * iv. Injectable
  * Progestogen-only hormonal contraception

    * v. Oral
    * vi. Injectable
  * Highly Effective Methods That Have Low User Dependency (Failure rate of <1% per year when used consistently and correctly)

    * Progestogen- only contraceptive implant
    * Intrauterine hormone-releasing system (IUS) Intrauterine device (IUD)
    * Bilateral tubal occlusion
    * Vasectomized partner (A vasectomized partner is a highly effective contraception method provided that the partner is the sole male sexual partner of the WOCBP and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used).
    * Sexual abstinence (Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant).
    * NOTES: Use should be consistent with local regulations regarding the use of contraceptive methods for participants of clinical studies.

      * a. Typical use failure rates are lower than perfect-use failure rates (i.e. when used consistently and correctly).
      * b. If hormonal contraception efficacy is potentially decreased due to interaction with study treatment, condoms must be used in addition to the hormonal contraception during the treatment period and for at least during study treatment and for 120 days after study treatment discontinuation after the last dose of study treatment or the initiation of other cancer therapy (whichever is shorter).
      * c. If locally required, in accordance with Clinical Trial Facilitation Group (CTFG) guidelines, acceptable contraceptive implants are limited to those which inhibit ovulation.
* Male participants must agree to use at least one of the following methods of contraception starting with the first dose of study therapy through 120 days after the last dose of therapy or the initiation of other cancer therapy (whichever is shorter):

  * Be abstinent from penile-vaginal intercourse as their usual and preferred lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent
  * Use a male condom plus partner use of a contraceptive method with a failure rate of <1% per year when having penile-vaginal intercourse with a woman of childbearing potential who is not currently pregnant.

    * a. Note: Men with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile penetration.

Exclusion Criteria:

* Received any therapy for tumor recurrence other than surgery;
* More than one episode of recurrent or progressive tumor;
* Is currently participating or plans to participate in another study of an investigational agent or using an investigational device.
* Tumor primarily localized to the brainstem or spinal cord;
* Presence of multifocal tumor, bi-hemispheric tumor (radiographic evidence of tumor extending from one hemisphere into the other through the corpus callosum), diffuse leptomeningeal or extracranial disease;
* Has a diagnosis of immunodeficiency;
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator. Examples include - but are not limited to - unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements;
* Has history of known coagulopathy that increases risk of bleeding or a history of clinically significant hemorrhage within 12 months of enrollment;
* Has evidence of intratumoral or peritumoral hemorrhage on baseline MRI scan other than those that are grade ≤ 1 and either post-operative or stable on at least 2 consecutive MRI scans;
* Has gastrointestinal bleeding or any other hemorrhage/bleeding event CTCAE Grade > 3 within 6 months of enrollment;
* Has a known additional malignancy that is progressing or requires active treatment within 1 year of start of study drug, except for those treated with surgical therapy only (e.g. basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy);
* Has active autoimmune disease requiring systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg thyroxine, insulin, or physiologic corticosteroid replacement for adrenal insufficiency or pituitary/hypothalamic dysfunction, etc.) is not considered a form of systemic treatment;
* Has history of (non-infectious) pneumonitis that required steroids or has current pneumonitis;
* Has an active infection requiring systemic therapy within 7 days before enrollment;
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial;
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) and is receiving antiretroviral therapy.
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected);
* Has a history of non-healing wounds or ulcers, or bone refractures within 3 months of fracture;
* Has a history of arterial thromboembolism within 12 months of enrollment;
* Has had clinically significant cardiovascular disease within 12 months of start of study drug, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure, or arrhythmias not controlled by outpatient medication, percutaneous transluminal coronary angioplasty/stent;
* Has a known history of active TB (Bacillus Tuberculosis);
* Has a known hypersensitivity to any of the study therapy products and/or any of their excipients;
* Is pregnant or breastfeeding or expecting to conceive within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment or the initiation of other cancer therapy (whichever is shorter). Pregnant women are excluded because there is an unknown but potential risk for adverse events affecting a developing fetus and/or the mother secondary to treatment with CUE-102. There is also an unknown but potential risk for adverse events affecting nursing infants secondary to treatment of the mother with CUE-102, thus, breastfeeding must be discontinued if the mother is treated with CUE-102;
* Is receiving any form of immunosuppressive therapy (e.g. chronic systemic steroid therapy exceeding dosage of 10 mg daily of prednisone equivalent) within 7 days prior to enrollment;
* Has received systemic immunosuppressive treatments, aside from systemic corticosteroids (such as methotrexate, chloroquine, azathioprine, etc), within six months of enrollment;
* Requires treatment with high dose systemic corticosteroids defined as dexamethasone > 2 mg/day or bioequivalent for at least 3 consecutive days within 2 weeks of enrollment;

  * Inhaled or topical steroids and adrenal replacement doses ≤ 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
  * Participants are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption).
  * Physiologic replacement doses of systemic corticosteroids are permitted, ≤10 mg/day prednisone equivalents.
  * A brief course of corticosteroids for prophylaxis (eg, contrast dye allergy) or for treatment of non-autoimmune conditions (eg, delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
* Requires therapeutic anticoagulation with warfarin at baseline; patients must be off warfarin or warfarin-derivative anti-coagulants for at least 7 days prior to enrollment; however, therapeutic or prophylactic therapy with low-molecular weight heparin is allowed;
* Has received a live vaccine within 30 days prior to enrollment;

  * Examples of live vaccines include - but are not limited to - the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette- Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* History of acute pancreatitis within 3 months before enrollment;
* Diverticulitis that is clinically significant in the opinion of the Investigator based on the extent or severity of known disease and/or the occurrence of clinically significant flares within 4 weeks before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose-limiting-toxicities (DLT) | 3 weeks
  A DLT is defined as any adverse event (AE) considered related to CUE-102 that meets DLT criteria in the 21-day period following the first dose of CUE-102 including pre-treatment laboratory results required for C2D1.
Maximum Tolerated Dose (MTD) | 3 weeks
  MTD is determined using a 3+3 design as listed in protocol section 1.1

SECONDARY OUTCOMES:
Safety and tolerability | Up to 1 year
  safety and tolerability as measured by CTCAEv5.0 including clinical, laboratory, EKG and radiographic assessments.

CONTACTS AND LOCATIONS:
Overall Officials: David Reardon, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu